CLINICAL TRIAL: NCT00537147
Title: Phase 1 Study of the Safety and Immunogenicity of a 2-Dose Regimen of West Nile/Dengue 4-3'delta30 Chimeric Virus Vaccine (WN/DEN4delta30), a Live Attenuated Vaccine for West Nile Encephalitis
Brief Title: Safety of and Immune Response to a West Nile Virus Vaccine (WN/DEN4delta30) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 242; WIRB Protocol Number 20071891
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: West Nile Fever
Keywords: Chimeric West Nile Virus; West Nile Virus; Dengue Virus
MeSH Terms: conditions — West Nile Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 1 vaccination of a 10^4 plaque-forming units (PFU) dose of WN/DEN4delta30 vaccine administered as 0.5 ml subcutaneously in deltoid at study entry and Day 180.
  Interventions: Biological: WN/DEN4delta30 vaccine
- 2 (Experimental): 1 vaccination of a 10^5 PFU dose of WN/DEN4delta30 vaccine administered as 0.5 ml subcutaneously in deltoid at study entry and Day 180.
  Interventions: Biological: WN/DEN4delta30 vaccine
- 3 (Placebo Comparator): 1 vaccination of a placebo administered as 0.5 ml subcutaneously in deltoid at study entry and Day 180.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: WN/DEN4delta30 vaccine — Live attenuated WN/DEN4delta30 vaccine (one of two doses)
  Arms: 1; 2
Biological: Placebo — Placebo for WN/DEN4delta30 vaccine
  Arms: 3

SUMMARY:
West Nile (WN) virus infection is an emerging disease. Infection with WN virus may lead to paralysis, coma, and death. The purpose of this study is to determine the safety of and immune response to a two-dose regimen of a WN vaccine in healthy adults. The vaccine is based on a live attenuated vaccine developed against dengue virus.

DETAILED DESCRIPTION:
WN is widely distributed in Africa and Europe, where it is usually associated with mild illness. In the United States, WN is considered a public health threat because severe illness caused by WN infection has caused paralysis, coma, and death, especially in the elderly. This study will evaluate the safety and immunogenicity of a live attenuated chimeric virus, WN/DEN4delta30, which is derived from the DEN4 dengue virus and wild-type WN serotypes.

This study will last at least 32 weeks. Participants in Cohort 1 will be randomly assigned to receive 1X10^4 plaque-forming units (PFU) WN/DEN4delta30 or placebo at study entry and Day 180. Cohort 2 will be randomly assigned to receive a higher dose of WN/DEN4delta30, 10^5 PFU, or placebo at study entry and Day 180. Immediately after receiving their injections, participants will be observed for 30 minutes for immediate adverse reactions.

After each vaccination, participants will be asked to monitor their temperatures three times every day for 16 days. Study visits will occur every other day after each vaccination until Day 16, followed by three additional visits at selected days through Day 180 post-vaccination. Blood collection, medical history, vital signs measurement, and a targeted physical exam will occur at all visits. Participants will also be required to keep temperature diaries until Day 16 after vaccination. Female participants will have a urine pregnancy test performed within 60 days of study entry, and on Days 28, 42, 150, 180, 208, and 222. Pregnancy prevention counseling will occur at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Available for the duration of the trial
* Willing to use acceptable forms of contraception for the duration of the study

Exclusion Criteria:

* Clinically significant neurologic, heart, lung, liver, rheumatologic, autoimmune, or kidney disease
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the ability of the volunteer to understand and cooperate with the study
* Neutropenia (abnormally low neutrophil count)
* Alcohol or drug abuse within 12 months prior to study entry
* Elevated levels of alanine aminotransferase (ALT) and serum creatinine
* History of severe allergic reaction or anaphylaxis
* Severe asthma
* HIV-1 infected
* Hepatitis C virus infected
* Hepatitis B surface antigen positive
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs within 30 days of study entry. Participants who have used topical or nasal corticosteroids are not excluded.
* Live vaccine within 4 weeks prior to study entry
* Killed vaccine within 2 weeks prior to study entry
* Surgical removal of spleen
* Blood products within 6 months prior to study entry
* History of dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis, West Nile virus)
* Previously received a licensed or experimental yellow fever or dengue vaccine
* Investigational agent within 30 days of study entry
* Other condition that, in the opinion of the investigator, would affect the participant's participation in the study
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related adverse events, as classified by both intensity and severity through active and passive surveillance | Throughout study
Immunogenicity, determined by anti-WN/DEN4 neutralizing antibody titer | At study entry, Days 28 and 42 after first vaccination, and Days 180, 208, and 222 after second vaccination

SECONDARY OUTCOMES:
Assess the frequency, quantity, and duration of viremia after each dose of vaccine by dose cohort (10^4 or 10^5 PFU) | Throughout study
Determine the number of vaccinees infected with WN/DEN4delta30 in each dose cohort (10^4 or 10^5 PFU) | Throughout study
Compare the infectivity rates, safety, and immunogenicity between dose 1 and dose 2 within a cohort and between cohorts | At study completion

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, M.D., Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research, Johns Hopkins School of Public Health (DC Location), Washington D.C., District of Columbia
  - Center for Immunization Research, Johns Hopkins School of Public Health (MD Location), Baltimore, Maryland

REFERENCES:
- [Background] Chang GJ, Kuno G, Purdy DE, Davis BS. Recent advancement in flavivirus vaccine development. Expert Rev Vaccines. 2004 Apr;3(2):199-220. doi: 10.1586/14760584.3.2.199. PMID 15056045
- [Background] Pletnev AG, Claire MS, Elkins R, Speicher J, Murphy BR, Chanock RM. Molecularly engineered live-attenuated chimeric West Nile/dengue virus vaccines protect rhesus monkeys from West Nile virus. Virology. 2003 Sep 15;314(1):190-5. doi: 10.1016/s0042-6822(03)00450-1. PMID 14517072